CLINICAL TRIAL: NCT00104507
Title: A 4-Week, Dose-ranging, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Assess the Safety and Efficacy of APD356 in Obese Patients
Brief Title: Safety and Efficacy of APD356 in the Treatment of Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APD356-003
Record Dates: First submitted 2005-03-01; First posted 2005-03-02 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2006-12

CONDITIONS: Obesity
Keywords: Serotonin; 5-HT2c; Satiety; Obesity; Appetite suppressant; Weight Loss; Overweight
MeSH Terms: conditions — Obesity; Anorexia; Weight Loss; Overweight | interventions — lorcaserin

INTERVENTIONS:
Drug: APD356

SUMMARY:
This is a research study of an investigational drug, APD356, a novel, selective 5-HT2c receptor agonist, in clinical development as a potential treatment for obesity.

The purpose of this study is to obtain preliminary assessment of the safety and efficacy of APD356, when administered daily for 28 days, in obese subjects who are otherwise healthy.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, randomized, parallel group study. Three different doses of APD356 or placebo will be administered daily for 28 days, to uncomplicated obese, male and nonpregnant, nonlactating, female volunteers, aged 18 to 65 years. Approximately 400 subjects will be enrolled.

ELIGIBILITY:
* Healthy male or nonpregnant, nonlactating females aged between 18 and 65 years (inclusive)
* Body Mass Index (BMI) of 30-45 Kg/m^2.
* Non-smoker
* No concomitant medications
* No past treatment with drugs associated with the development of pulmonary hypertension or cardiac valvular insufficiency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2004-12 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Change in body weight

SECONDARY OUTCOMES:
Safety
Changes in waist circumference, hip circumference and waist/hip ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- See also: obesity information — http://obesity.org/
- See also: N. American Association for the Study of Obesity web page — http://www.obesity.org/
- See also: sponsor company web page — http://www.arenapharm.com
- See also: Pennington Biomedical Research Center home web page — http://www.pbrc.edu